CLINICAL TRIAL: NCT03478683
Title: A Phase IV, 12-week, Randomised, Double-blind, Triple Dummy Study to Compare Single Inhaler Triple Therapy, Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI) With Multiple Inhaler Therapy (Budesonide/Formoterol Plus Tiotropium) Based on Lung Function and Symptoms in Participants With Chronic Obstructive Pulmonary Disease
Brief Title: A Randomized Study, Comparing Fluticasone Furoate/Umeclidinium/Vilanterol (FF/UMEC/VI) Single Inhaler Triple Therapy, Versus Multiple Inhaler Therapy (Budesonide/Formoterol Plus Tiotropium) in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207608; 2017-001149-28 (EudraCT Number)
Record Dates: First submitted 2018-03-23; First posted 2018-03-27 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: long-acting muscarinic receptor antagonists; tiotropium; HRQoL; Budesonide/formoterol; chronic obstructive pulmonary disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Albuterol; Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: This is a parallel group study. Eligible subjects will be randomized in a ratio of 1:1 to receive either FF/UMEC/VI single inhaler triple therapy or multiple inhaler triple combination therapy (budesonide/formoterol plus tiotropium) during the treatment period.
Who Masked: Participant, Investigator
Masking Description: This is a phase 4 double blind study, which will use a triple dummy design for dosing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- FF/UMEC/VI 100/62.5/25 mcg (Experimental): Subjects will receive budesonide/formoterol (320/9 mcg) twice daily plus tiotropium (18 mcg) once daily plus placebo via ELLIPTA during the 4-week run-in period. Subjects will be administered FF/UMEC/VI 100/62.5/25 mcg via ELLIPTA once daily in the morning plus placebo to match budesonide/formoterol via MDI, two inhalations twice daily plus placebo to match tiotropium via HandiHaler once daily in the morning for 84 days in the treatment period.
  Interventions: Drug: budesonide/formoterol; Drug: albuterol/salbutamol; Drug: FF/UMEC/VI; Drug: Placebo to match budesonide/formoterol; Drug: tiotropium; Drug: placebo to match tiotropium; Device: ELLIPTA; Device: MDI; Device: HandiHaler
- Budesonide/formoterol plus tiotropium (Active Comparator): Subjects will receive budesonide/formoterol (320/9 mcg) twice daily plus tiotropium (18 mcg) once daily plus placebo via ELLIPTA during the 4-week run-in period. Subjects will be administered budesonide/formoterol 160/4.5 mcg via MDI, two inhalations twice daily plus tiotropium 18 mcg via HandiHaler once daily in the morning plus placebo via ELLIPTA once daily in the morning for 84 days in the treatment period.
  Interventions: Drug: budesonide/formoterol; Drug: albuterol/salbutamol; Drug: tiotropium; Drug: Placebo to match FF/UMEC/VI; Device: ELLIPTA; Device: MDI; Device: HandiHaler

INTERVENTIONS:
Drug: budesonide/formoterol — Subjects will be administered two inhalations of budesonide/formoterol via MDI twice daily
Drug: albuterol/salbutamol — Subjects will be provided short-acting albuterol/salbutamol as-rescue medication to be used on an as-needed basis throughout the study.
Drug: FF/UMEC/VI — Subjects will receive FF/UMEC/VI 100/62.5/25 mcg via ELLIPTA once daily in the morning
  Arms: FF/UMEC/VI 100/62.5/25 mcg
Drug: Placebo to match budesonide/formoterol — Subjects will be administered two inhalations of matching placebo twice daily via MDI
  Arms: FF/UMEC/VI 100/62.5/25 mcg
Drug: tiotropium — Subjects will receive tiotropium (18 mcg) once daily in the morning via HandiHaler device
Drug: Placebo to match FF/UMEC/VI — Matching placebo to FF/UMEC/VI will be administered via ELLIPTA once daily in the morning.
  Arms: Budesonide/formoterol plus tiotropium
Drug: placebo to match tiotropium — Subjects will receive tiotropium matching placebo via Handihaler once daily in the morning
  Arms: FF/UMEC/VI 100/62.5/25 mcg
Device: ELLIPTA — Subjects will receive FF/UMEC/VI 100/62.5/25 mcg and matching placebo via ELLIPTA in the treatment period. Budesonide/formoterol plus tiotropium once daily plus placebo will be administered via ELLIPTA during the run-in period.
Device: MDI — Subjects will receive budesonide/formoterol and placebo to match budesonide/formoterol via MDI in the treatment period.
Device: HandiHaler — Subjects will be administered tiotropium (18 mcg) or placebo to match tiotropium via HandiHaler during the treatment period.

SUMMARY:
The primary purpose of this study is to evaluate lung function and health related quality of life (HRQoL) after 84 days of treatment with a single inhaler triple therapy combination of FF/UMEC/VI [100/62.5/25 microgram (mcg)] once daily via the ELLIPTA™ compared with a multiple inhaler combination therapy of Symbicort Metered Dose Inhaler (MDI) (budesonide/formoterol 320/9 mcg) twice daily plus Spiriva HandiHaler (tiotropium 18 mcg) once daily. The study will inform healthcare providers that subjects can be effectively and safely switched to FF/UMEC/VI single inhaler therapy from a multiple inhaler triple therapy regimen of Symbicort MDI and Spiriva Handihaler. Eligible subjects will enter a 4-week run-in period during which they will be administered budesonide/formoterol (320/9 mcg) twice daily plus tiotropium (18 mcg) once daily plus placebo via ELLIPTA. Following the run-in period, subjects will be randomized to receive one of the following study treatments for 84 days: 1) FF/UMEC/VI 100/62.5/25 mcg via ELLIPTA once daily in the morning plus two inhalations of placebo to match budesonide/formoterol via MDI, twice daily plus placebo to match tiotropium via HandiHaler once daily in the morning or 2) Budesonide/formoterol 320/9 mcg via MDI, twice daily plus tiotropium 18 mcg via HandiHaler once daily in the morning plus placebo via ELLIPTA once daily in the morning. Subjects will then enter a one week follow-up period. The total duration for a subject in the study will be approximately 17 weeks. ELLIPTA is a registered trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be capable of giving signed informed consent prior to study start.
* Only outpatient subjects will be included
* Subjects (male or female) must be 40 years of age or older at Screening (Visit 1). A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and until safety follow-up contact after the last dose of study treatment
* An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society
* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years at Screening (Visit 1) [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* Subjects with a score of >=10 on the COPD Assessment Test (CAT) at Screening (Visit 1)
* Subjects must demonstrate a post-bronchodilator FEV1 <50 % predicted normal or a post-bronchodilator FEV1 <80 % predicted normal and a documented history of >=2 moderate exacerbations or one severe (hospitalized) exacerbation in the previous 12 months. Subjects must also have a measured post albuterol/salbutamol FEV1/forced vital capacity (FVC) ratio of <0.70 at screening
* Subjects must have been receiving daily maintenance treatment for their COPD for at least 3 months prior to Screening

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study
* Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD).
* Subjects with alpha 1-antitrypsin deficiency as the underlying cause of COPD
* Subjects with active tuberculosis, lung cancer, and clinically significant: bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung disease or other active pulmonary diseases
* Subjects who have undergone lung volume reduction surgery within the 12 months prior to Screening
* Immune suppression (e.g. advanced human immunodeficiency virus [HIV] with high viral load and low cluster of differentiation 4 [CD4] count, lupus on immunosuppressants) that in the opinion of the investigator would increase risk of pneumonia or other risk factors for pneumonia (e.g. neurological disorders affecting control of the upper airway, such as Parkinson's Disease, Myasthenia Gravis).
* Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening and at least 30 days following the last dose of oral or systemic corticosteroids (if applicable)
* Respiratory tract infection that has not resolved at least 7 days prior to Screening
* Chest x-ray (posteroanterior and lateral) reveals evidence of pneumonia or a clinically significant abnormality not believed to be due to the presence of COPD, or another condition that would hinder the ability to detect an infiltrate on chest X-ray (e.g. significant cardiomegaly, pleural effusion or scarring). All subjects will have a chest X-ray at Screening Visit 1 (or historical radiograph or computerized tomography [CT] scan obtained within 3 months prior to screening). For sites in Germany: If a chest x-ray (or CT scan) within 3 months prior to Screening (Visit 1) is not available, approval to conduct a diagnostic chest x-ray will need to be obtained from the Federal Office for Radiation Protection (BfS).
* Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Unstable liver disease: alanine transaminase (ALT) >2 times Upper Limit of Normal (ULN); and bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 %). Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Subjects with any of the following at Screening (Visit 1) would be excluded: Myocardial infarction or unstable angina in the last 6 months; Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months; New York Heart Association (NYHA) Class IV Heart failure.
* Abnormal and clinically significant 12-lead electrocardiogram (ECG) finding at Visit 1. The Investigator will determine the clinical significance of each abnormal ECG finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial. An abnormal and clinically significant finding that would preclude a subject from entering the trial is defined as a 12-lead ECG tracing that is interpreted at, but not limited to, any of the following: i) Atrial Fibrillation (AF) with rapid ventricular rate >120 beats per minute (BPM); ii) Sustained and non-sustained Ventricular tachycardia (VT); iii). Second degree heart block Mobitz type II and third degree heart block (unless pacemaker or defibrillator had been inserted); iv) QT interval corrected for heart rate by Fridericia's formula (QTcF) >=500 milliseconds (msec) in subjects with QRS <120 msec and QTcF >=530 msec in subjects with QRS >=120 msec.
* A history of allergy or hypersensitivity to any corticosteroid, anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the Investigator, contraindicates study participation.
* Subjects with carcinoma that has not been in complete remission for at least 3 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 3 year waiting period if the subject has been considered cured by treatment.
* Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3 liters per minute (L/min) at screening (Oxygen use <=3 L/min flow is not exclusionary)
* Subjects who are medically unable to withhold their albuterol/salbutamol for the 4-hour period required prior to spirometry testing at each study visit
* Subjects who have participated in the acute phase of a Pulmonary Rehabilitation Programme within 4 weeks prior to screening or subjects who plan to enter the acute phase of a Pulmonary Rehabilitation Program during the study. Subjects who are in the maintenance phase of a Pulmonary Rehabilitation Program are not excluded.
* Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years
* Subjects at risk of non-compliance, or unable to comply with the study procedures. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study
* Study Investigators, sub-Investigators, coordinators, employees of a participating Investigator or study site, or immediate family members of the aforementioned that is involved with this study
* In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete study related materials
* Use of various medication prior to screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (50):
- United States (34):
  - GSK Investigational Site, Gold River, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeBary, Florida
  - GSK Investigational Site, Edgewater, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Peachtree Corners, Georgia
  - GSK Investigational Site, Flint, Michigan
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Woodbury, Minnesota
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Fort Mill, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Lancaster, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Baytown, Texas
  - GSK Investigational Site, Cypress, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Tomball, Texas
- Czechia (5):
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kralupy nad Vltavou
  - GSK Investigational Site, Lovosice
  - GSK Investigational Site, Rokycany
  - GSK Investigational Site, Teplice
- Germany (6):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Netherlands (5):
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Heerlen
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Zutphen

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20594

REFERENCES:
- [Background] Ferguson GT, Brown N, Compton C, Corbridge TC, Dorais K, Fogarty C, Harvey C, Kaisermann MC, Lipson DA, Martin N, Sciurba F, Stiegler M, Zhu CQ, Bernstein D. Once-daily single-inhaler versus twice-daily multiple-inhaler triple therapy in patients with COPD: lung function and health status results from two replicate randomized controlled trials. Respir Res. 2020 May 29;21(1):131. doi: 10.1186/s12931-020-01360-w. PMID 32471423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, multicenter, parallel group study where participants with chronic obstructive pulmonary disease (COPD) were randomized to receive either fluticasone furoate/umeclidinium/vilanterol or budesonide/formoterol plus tiotropium in a 1:1 ratio. The study was conducted across 65 centers in 4 countries.
Pre-assignment Details: A total of 1036 participants were screened in the study, of which 215 failed during screening. Of the 821 participants who entered the run-in period, 92 were run-in failures. A total of 729 participants were randomized in the study, of which one participant was randomized in error. A total of 728 participants received randomized treatment.
Groups:
- Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg: Participants received fluticasone furoate/umeclidinium/vilanterol (FF/UMEC/VI) 100/62.5/25 microgram (mcg) via the ELLIPTA (once daily in the morning) plus placebo to match budesonide/formoterol (BUD/FOR) via metered dose inhaler (MDI) (two inhalations twice daily) plus placebo to match tiotropium (TIO) via HandiHaler (once daily in the morning) for 84 days. Participants received albuterol/salbutamol as rescue medication during conduct of the study, if required.
- Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg: Participants received two inhalations of budesonide/formoterol 160/4.5 mcg via MDI in the morning and two inhalations in the evening (total dose of 320/9 mcg twice daily) plus tiotropium 18 mcg via HandiHaler (once daily in the morning) plus placebo to match fluticasone furoate/umeclidinium/vilanterol via the ELLIPTA (once daily in the morning) for 84 days. Participants received albuterol/salbutamol as rescue medication during conduct of the study, if required.
Period: Overall Study
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg
Started | 363 | 365
Completed | 350 | 347
Not Completed | 13 | 18
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 0 | 5
Not completed — Physician Decision | 1 | 3
Not completed — Withdrawal by Subject | 7 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants, excluding those who were randomized in error.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg | Total
Number analyzed (Participants) | 363 | 365 | 728
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (7.90) | 64.9 (8.06) | 65.2 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 164 | 344
  Male | 183 | 201 | 384
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 34 | 33 | 67
  American Indian Or Alaska Native | 0 | 1 | 1
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  Asian - South East Asian Heritage | 0 | 1 | 1
  White - Arabic/North African Heritage | 0 | 2 | 2
  White - White/Caucasian/European | 327 | 328 | 655
  Multiple | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) Over 0-24 Hours at Week 12 for Modified Per Protocol (mPP) Population
Description: FEV1 is an important measure of pulmonary function and is the maximum amount of air that can be forced out in one second after taking a deep breath. FEV1 was measured using spirometry. Serial FEV1 assessments were performed at multiple time points (-30 and -5 minutes pre-dose, and 5 minutes, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 12 hours, 15 hours, 21 hours, 23 hours and 24 hours post-dose) over 24-hour period at Week 12. Weighted mean change from Baseline at week 12 was calculated by subtracting weighted mean FEV1 at week 12 from Baseline FEV1, where Baseline FEV1 is the average of the two FEV1 measurements made at 30 minutes and 5 minutes pre-dose on Day 1. The weighted mean was derived by calculating the area under the FEV1 time curve (AUC) over the actual time of assessment relative to the time of dosing (over 24-hour period) using the trapezoidal rule, and then dividing the value by the time interval (24-hour) over which the AUC was calculated.
Time Frame: Baseline and Week 12
Population: mPP Population comprised of all participants in the ITT population who do not have a protocol deviation of not meeting eligibility criteria or not meeting randomization criteria. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg
Number analyzed (Participants) | 282 | 272
Liters | 0.045 (0.0101) | 0.030 (0.0101)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg; Test type: Non-Inferiority — Non-inferiority was to be demonstrated, if the lower bound of the two-sided 95 percentage (%) confidence interval around the (FF/UMEC/VI versus BUD/FOR+TIO) treatment difference was above -50 milliliter; Mean Difference (Net) = 0.015, 95% CI 2-sided [-0.013 to 0.043], Standard Error of Mean 0.0143 — The primary treatment effect estimated (hypothetical effect) excluded data following intercurrent events: discontinuation of treatment, taking wrong treatment, taking prohibited medication, unblinding, noncompliance, COPD exacerbation or pneumonia

2. Secondary Outcome: Change From Baseline in Trough FEV1 on Day 2, Day 28, Day 84 and Day 85
Description: FEV1 is an important measure of pulmonary function and is the maximum amount of air that can be forced out in one second after taking a deep breath. FEV1 was measured using spirometry. For Day 2 and Day 85, trough FEV1 was defined as the mean of the 23-hour and 24-hour serial spirometry FEV1 measurements. For Day 28 and Day 84, trough FEV1 was defined as the average of the pre-dose FEV1 measurements recorded before the morning dose of randomized study treatment. Change from Baseline in trough FEV1 was calculated by subtracting post-dose trough FEV1 value from Baseline FEV1, where Baseline FEV1 is the average of the two FEV1 measurements made at 30 minutes and 5 minutes pre-dose on Day 1. The treatment effect to be estimated for trough FEV1 was hypothetical effect if all participants stayed on their randomized study treatment. Only on treatment data was included in analysis.
Time Frame: Baseline, Days 2, 28, 84 and 85
Population: ITT Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg
Number analyzed (Participants) | 358 | 359
Liters
  Day 2, n=358,359 | 0.008 (0.0098) | 0.018 (0.0098)
  Day 28, n=355,353: number analyzed (Participants) | 355 | 353
  Day 28, n=355,353 | 0.046 (0.0088) | -0.015 (0.0088)
  Day 84, n=344,340: number analyzed (Participants) | 344 | 340
  Day 84, n=344,340 | 0.040 (0.0094) | -0.018 (0.0094)
  Day 85, n=341,337: number analyzed (Participants) | 341 | 337
  Day 85, n=341,337 | 0.026 (0.0099) | -0.012 (0.0099)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg; Test type: Superiority; p = 0.481, Mixed model repeated measures — Only if superiority is achieved on the primary study endpoint, then inferences can be made on change from Baseline in trough FEV1 on Day 2 using p-values; Mean Difference (Net) = -0.010, 95% CI 2-sided [-0.037 to 0.018], Standard Error of Mean 0.0139 — Day 2
Statistical Analysis 2: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg; Test type: Superiority; p < 0.001, Mixed model repeated measures — Only if superiority is achieved on the primary study endpoint, then inferences can be made on change from Baseline in trough FEV1 on Day 28 using p-values; Mean Difference (Net) = 0.061, 95% CI 2-sided [0.037 to 0.086], Standard Error of Mean 0.0124 — Day 28
Statistical Analysis 3: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg; Test type: Superiority; p < 0.001, Mixed model repeated measures — Only if superiority is achieved on the primary study endpoint, then inferences can be made on change from Baseline in trough FEV1 on Day 84 using p-values; Mean Difference (Net) = 0.058, 95% CI 2-sided [0.032 to 0.084], Standard Error of Mean 0.0133 — Day 84
Statistical Analysis 4: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg; Test type: Superiority; p = 0.007, Mixed model repeated measures — Only if superiority is achieved on the primary study endpoint, then inferences can be made on change from Baseline in trough FEV1 on Day 85 using p-values; Mean Difference (Net) = 0.038, 95% CI 2-sided [0.010 to 0.066], Standard Error of Mean 0.0140 — Day 85

3. Secondary Outcome: Weighted Mean Change From Baseline in FEV1 Over 0-24 Hours on Day 1
Description: FEV1 is an important measure of pulmonary function and is the maximum amount of air that can be forced out in one second after taking a deep breath. FEV1 was measured using spirometry. Serial FEV1 assessments were performed at multiple time points (-30 and -5 minutes pre-dose, and 5 minutes, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 12 hours, 15 hours, 21 hours, 23 hours and 24 hours post-dose) over 24-hour period on Day 1. Weighted mean change from Baseline on Day 1 was calculated by subtracting weighted mean FEV1 on Day 1 from Baseline FEV1, where Baseline FEV1 is the average of the two FEV1 measurements made at 30 minutes and 5 minutes pre-dose on Day 1. The weighted mean was derived by calculating the area under the FEV1 time curve (AUC) over the actual time of assessment relative to the time of dosing (over 24-hour period) using the trapezoidal rule, and then dividing the value by the time interval (24-hour) over which the AUC was calculated.
Time Frame: Baseline and Day 1
Population: ITT Population. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg
Number analyzed (Participants) | 354 | 355
Liters | 0.054 (0.0078) | 0.063 (0.0077)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg; Test type: Superiority; p = 0.415, Mixed model repeated measures — Only if superiority is achieved on the primary study endpoint, then inferences can be made on weighted mean change from Baseline in FEV1 over 0-24 hours on Day 1 using p-values; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.030 to 0.013], Standard Error of Mean 0.0110 — The treatment effect to be estimated was hypothetical effect if all participants stayed on their randomized study treatment. Only on treatment data was included in analysis

4. Primary Outcome: Weighted Mean Change From Baseline in FEV1 Over 0-24 Hours at Week 12 for ITT Population
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: ITT Population comprised of all randomized participants, excluding those who were randomized in error. Only those participants with data available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg
Number analyzed (Participants) | 336 | 332
Liters | 0.046 (0.0097) | 0.032 (0.0098)
Statistical Analysis 1: Comparison: Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg vs Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg; Test type: Superiority; p = 0.335, Mixed model repeated measures — The analysis was performed using mixed model repeated measures analysis, which included covariates of Baseline FEV1, geographical region, treatment, visit, visit by treatment and visit by Baseline interaction; Mean Difference (Net) = 0.013, 95% CI 2-sided [-0.014 to 0.040], Standard Error of Mean 0.0138 — [estimate comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were reported from start of study treatment and up to Week 13
Description: Non-SAEs and SAEs were reported for ITT Population. Adverse events were presented treatment-wise.
Arm/Group | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg
All-Cause Mortality (participants affected / at risk) | 0/363 | 0/365
Serious Adverse Events (participants affected / at risk) | 29/363 | 16/365
Other Adverse Events (participants affected / at risk) | 18/363 | 12/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg (N=363) | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg (N=365)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Psoas abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Furoate/Umeclidinium/Vilanterol 100/62.5/25 mcg (N=363) | Budesonide/Formoterol 320/9 mcg Plus Tiotropium 18 mcg (N=365)
Nasopharyngitis (Infections and infestations) | 18 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03478683/SAP_000.pdf
  • Study Protocol (2018-07-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT03478683/Prot_001.pdf